CLINICAL TRIAL: NCT03920059
Title: A Randomized Open-label Study of Fixed-dose Versus Concentration-controlled Mycophenolate Mofetil for the Treatment of Active Lupus Nephritis
Brief Title: Fixed-dose Versus Concentration-controlled Mycophenolate Mofetil for the Treatment of Active Lupus Nephritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Chulalongkorn University (Other)
Collaborators: Berlin Pharmaceutical Industry (Unknown)
Responsible Party: Principal Investigator, Yingyos Avihingsanon, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDCC lupus
Record Dates: First submitted 2019-04-01; First posted 2019-04-18 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FD arm (Placebo Comparator): MMF will be prescribed at a starting dose of 1.5 g/day and increased to 2 g/day at week 4 (if body weight ≥ 45 kg) and continue the same dose until week 24. After week 24, MMF will be lowered to 1.5 g/day.
  Interventions: Drug: Mycophenolate Mofetil
- CC Arm (Active Comparator): MMF will be prescribed at a starting dose of 1.5 g/day. MPA-C0 (trough) level will be measured weekly and MMF dose will be increased by 500 mg/day every week until the MPA-C0 level ≥ 3 mg/L or the MMF dosage is 3000 mg/day. After achieving the targeted MPA-C0 level, the MMF dose adjustment will be allowed only if the MPA-C0 levels are lower than 3 mg/L for two consecutive monitoring visits. After week 12, MMF will be maintained at the same dose until week 48
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Description Each capsule contains Mycophenolate mofetil 250 mg. Presentation / Packing Cap 250 mg (white to off white powder, light blue/peach hard gelatin, imprinting with "MMF" on cap and "250" on body) x 10 x 10's.
  Storage Store below 30 degree Celcius.

SUMMARY:
A randomized open-label study of fixed-dose versus concentration-controlled mycophenolate mofetil for treatment of active lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 year
* Diagnosis of SLE according to ACR criteria. At least 4 criteria must have been present for the diagnosis of SLE
* Active lupus nephritis (both new and flare patients can be included) defined as:

  * Within 16 weeks of randomization, had Biopsy-proven ISN class III or IV [exclude III(c), IV-S(c) and IV-G(c). Patients are permitted to have co-existing class V and
  * At screening day, has urine protein creatinine ratio (UPCR) or 24-hour urinary protein ≥ 1.0 g/g or g/day

Exclusion Criteria:

* Pregnancy or breast feeding
* Child-bearing age women who refuse to use effective birth-control
* Poor compliance
* Estimated-GFR < 20 mL/min/1.73 m2
* Crescentic glomeruli more than 30 percent
* Severe extra-renal involvement of SLE
* History of severe allergic reactions or adverse effects to MMF
* Uncontrolled concomitant disease
* Known active, clinically significant infection of any kind
* History of serious recurrent or chronic infection
* History of malignancy (except basal cell carcinoma, squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been excised and cured)
* Concomitant conditions which has required treatment with systemic corticosteroid (excluding topical or inhaled steroids) at any time in the 52 weeks prior to screening
* Treatment with more than 1 g cyclophosphamide within the past 24 weeks
* Receipt more than 3 g of IV pulse methylprednisolone within the past 12 weeks
* Receipt prednisolone more than 30 mg/day for longer than 30 days within the past 12 weeks
* Treatment with MMF at ≥ 1.5 g/day for over 4 weeks within the past 12 weeks
* On treatment with Tacrolimus or Cyclosporine on the day of screening
* Treatment with any biologic B-cell depleting therapy (e.g. anti CD-20, anti CD 22) within 52 weeks
* Receiving concomitant medication interfering PK of MPA

  * Cholestyramine
  * Rifampin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Response rate at 48 week of therapy | 48 weeks

SECONDARY OUTCOMES:
Adverse events | 48 weeks
Mycophenolic acid trough levels | 48 weeks
MPA-area under the curve (AUC) 0-4 hour at 12 week | 12 weeks
C3 levels | 48 weeks
Urine IP-10 levels | 48 weeks
Anti-dsDNA | 48 weeks
Relapse free survival at 96, 144 and 240 week | 96, 144 and 240 weeks
eGFR at 96, 144 and 240 week | 96, 144 and 240 weeks
Progression to CKD stage 3 or more at 96, 144 and 240 week | 96, 144 and 240 weeks
End stage renal disease at 96, 144 and 240 week | 96, 144 and 240 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Please Select, Thailand